CLINICAL TRIAL: NCT03657485
Title: Probiotic Supplementation in the Term Newborns Delivered by Caesarean Section: a Randomized, Prospective Clinical Trials
Brief Title: Probiotic Supplementation in the Term Newborns Delivered by Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Joanna Hurkała, PhD MD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KBET/46/B/2014
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Microbiota, Cesarean Section, Probiotics, Dysbiosis
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Intervention Model Description: The patients we recruited were randomized into 2 groups- interventional or control group. For comparison we examined the stool samples of 32 healthy newborns delivered vaginally
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- interventional (Experimental): In the interventional group we supplemented the probiotic containing Bifidobacterium breve PB04 i Lactobacillus rhamnosus KL53A (FFbaby, IBSS Biomed SA, Poland) orally during the first hour of life and after 12 hours in mother's milk or formula (the total amount of the probiotic was 2 x 10 6 CFU bacteria).
  Interventions: Dietary Supplement: containing Bifidobacterium breve PB04, Lactobacillus rhamnosus KL53A
- control (No Intervention): No intervention. Feeding with mother milk
- comperative (No Intervention): Comparing stool composition of vaginally born newborns

INTERVENTIONS:
Dietary Supplement: containing Bifidobacterium breve PB04, Lactobacillus rhamnosus KL53A — we supplemented the probiotic orally during the first hour of life and after 12 hours in mother's milk or formula (the total amount of the probiotic was 2 x 10 6 CFU bacteria).
  Other Names: FFBaby
  Arms: interventional

SUMMARY:
Objectives: The gut microbiota plays pivotal role in the maintenance of human health. There are numerous factors, including the mode of delivery, that impact early gut colonization. Recent research focuses on probiotics' use in prophylaxy of gut dysbiosis in the newborns delivered by CS. We aimed to investigate whether a probiotic supplement in the newborns delivered by CS alter the pattern of gut colonization and has effect on decreasing risk of dysbiosis.

Methods: a prospective, randomized trial with a control group. 150 newborns, born in 38-40 gestational age, delivered by CS were included to the study. They were randomized into 2 groups- interventional supplemented with the probiotic containing Bifidobacterium breve PB04 i Lactobacillus rhamnosus KL53A (FFBaby, IBSS BioMed SA, Poland) and control. Stool samples were obtained on 5th and 6th day of life and after one month of life, and analyzed microbiologically in the lab. Bacterial colonies' genre and species were next identified and quantified.

DETAILED DESCRIPTION:
The aim of the study was to assess the effect of the probiotic supplementation on microbiota composition of the gut in healthy newborns delivered by CS. We studied colonization of GI tract on the day of discharge from hospital and after a month of life.

It was a prospective, randomized trial with the control group, conducted in the Neonatal Clinic of the Jagiellonian University Hospital in Kraków, lasting from April 2014 to April 2017.

The patients we recruited were randomized into 2 groups- interventional or control group. In the interventional group we supplemented the probiotic containing Bifidobacterium breve PB04 i Lactobacillus rhamnosus KL53A (FFBaby, IBSS BioMed SA, Poland) orally during the first hour of life and after 12 hours in mother's milk or formula (the total amount of the probiotic was 2 x 10 6 CFU bacteria).

The permission for the clinical trial was granted by the regional medical Bioethical Committee of the Jagiellonian University. (The number of decision- KBET/46/B/2014 from the 27th of March 2014)

ELIGIBILITY:
Inclusion Criteria:38-40 gestational age, normal, healthy pregnancy, delivery by CS, good clinical condition after birth, Apgar scale- 8-10 points, proper gestational mass> 2500g, informed consent of parents.

-

Exclusion Criteria:conditions mentioned above were not fulfilled, lack of informed consent of the parents or their resignation from the study.

-

Ages: 1 Hour to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
microbiota colonization | 1 month of life
  Stool microbiotic composition

SECONDARY OUTCOMES:
respiratory infection, gastrointestinal infection | 1 year of life
  frequency of respiratory and gastrointestinal infection

OTHER OUTCOMES:
allergy, atopy | 1 year of life
  allergy or atopy episodes

IPD SHARING:
Plan to Share IPD: No
participant data available for study statistics and laboratory stuff